CLINICAL TRIAL: NCT00173563
Title: Induction of Cytokines in Human Monocytes by SARS-CoV in Adults and Children
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Collaborators: National Science and Technology Council, Taiwan (Other Government)
Other Study IDs: 9461700731; NSC92-2751-B-002-026-Y
Record Dates: First submitted 2005-09-12; First posted 2005-09-15 (Estimated); Last update posted 2007-12-03 (Estimated); Status verified 2005-08

CONDITIONS: Healthy
Keywords: Immunology

STUDY DESIGN:
Time Perspective: Prospective

SUMMARY:
Severe acute respiratory syndrome (SARS) is a new emerging infectious disease. Its pathogen is a newly discovered coronavirus (SARS-CoV). The clinical course can be classified to 3 stages: viral replication phase, hyperimmune reactive phase, and pulmonary destruction phase. Human monocyte plays a critical role in the initiation of immune response in defending the intracellular pathogens (eg viruses). Monocytes can engulf viruses and present the viral antigens in the major histocompatibility (MHC) molecule to the cell surface to initiate T lymphocyte response. Monocytes also secrete various cytokines to modulate immune response. SARS-CoV is a mutant of animal virus to cause human disease and is able to cause unusual severe respiratory illness. It is suggested the unusual severe disease is due to the intense immune reaction.

The investigators will harvest human monocytes from healthy adult and children blood donors. Monocytes would be cultured and infected by SARS-CoV. The change of viral load is monitored after infection. Cytokines secreted by monocytes after infection are also measured. The difference of monocyte cytokine secretion is compared between adults and children. The study is to verify the SARS-CoV infectivity of human monocytes and prove the unusual severity caused by SARS-CoV is related to viral-induced dysregulation of cytokine responses. The results may also clarify why adults tend to have a more severe illness compared with children.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adults aged 20 to 50 years old
* Healthy children aged 2 to 5 years old

Ages: 2 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 10 (Estimated)
Dates: Start 2005-01; Study Completion 2005-09 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Luan-Yin Chang, MD, PhD, Principal Investigator — Department of pediatrics, National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan